CLINICAL TRIAL: NCT03605667
Title: A Phase 2 Randomized Double-Blind Placebo-Controlled Trial to Evaluate the Efficacy and Safety of BHV-4157 in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Study of BHV-4157 in Alzheimer's Disease
Acronym: T2 Protect AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biohaven Pharmaceuticals, Inc. (Industry)
Collaborators: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV4157-203
Record Dates: First submitted 2018-07-23; First posted 2018-07-30 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BHV-4157 (Experimental): troriluzole, 280 mg (2 x 140 mg) capsules, QD
  Interventions: Drug: troriluzole
- Placebo (Placebo Comparator): matching 280 mg (2 x 140 mg) placebo capsules, QD
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: troriluzole — Oral BHV-4157 will be given daily for up to 48 weeks
  Other Names: BHV-4157
  Arms: BHV-4157
Drug: Placebo oral capsule — Oral matching placebo will be given daily for up to 48 weeks
  Arms: Placebo

SUMMARY:
Preclinical models suggest that riluzole, the active metabolite of BHV-4157, may protect from AD-related pathology and cognitive dysfunction. Titrated dose of BHV-4157 to 280 mg, or placebo, were administered orally once daily. Duration of treatment is 48 weeks in double-blind phase. There is also a screening period of up to 42 days; and a 4-week post-treatment observation period. Eligible participants who completed the double-blind treatment phase had the opportunity to receive open-label troriluzole for up to 48 weeks in an open-label extension (OLE) phase.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 50 to 85 (inclusive) at screening
* Diagnosed with probable Alzheimer's disease dementia: Core clinical criteria in accordance with NIA/Alzheimer's Association Guidelines.
* Living in the community (includes assisted living facilities, but excludes long-term care nursing facilities).
* Ambulatory, or able to walk with an assistive device, such as a cane or walker.
* Participants must have a study partner who has frequent interaction with them (approximately >3-4 times per week), will be present for all clinic visits, and can assist in compliance with study procedures.
* An Mini-Mental State Examination score of 14 to 24, inclusive, at screening.
* A brain MRI scan within 6 months of screening consistent with a diagnosis of Alzheimer's disease.
* Participants should be treated with a stable dosage regimen of FDA-approved AD medications (acetylcholinesterase inhibitors (AchEI) and/or memantine) for at least 3 months prior to screening. Participants should be expected to remain on a stable dosage regimen of these medications for the duration of the trial.
* Participants who are not being treated with FDA-approved AD medications at the time of screening, because they have contraindications to these medications, or because they have previously failed treatment with these medications, are also eligible for inclusion, if it is expected that they will not be treated with these medications for the duration of the trial.

Key Exclusion Criteria:

* Hepatic impairment defined as Child-Pugh class of A or more severe liver impairment.
* Other neurodegenerative diseases and causes of dementias, including Parkinson's disease and Huntington's disease, vascular dementia, CJD (Creutzfeldt-Jakob disease), LBD (Lewy Body dementia), PSP (Progressive Supranuclear Palsy), AIDS (Acquired Immunodeficiency Syndrome), or NPH (normal pressure hydrocephalus).
* History of a major depressive episode within the past 6 months of screening.
* Insulin-dependent diabetes or uncontrolled diabetes with HbA1c value >8.0 %.
* Cancer or a malignant tumor within the past 3 years, except patients who underwent potentially curative therapy with no evidence of recurrence for >3 years. Patients with stable prostate cancer or non-melanoma skin cancers are not excluded.
* Participation in another clinical trial for an investigational agent and having taken at least one dose of study medication, unless confirmed as having been on placebo, within 12 weeks prior to screening. The end of a previous investigational trial is defined as the date of the last dose of an investigational agent.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-12-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - Xenoscience, Inc., Phoenix, Arizona
  - Barrow Neurological Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Neurology Center of North Orange County, Fullerton, California
  - University of California, San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - SC3 Research Group - Pasadena, Pasadena, California
  - Geriatric and Adult Psychiatry, Hamden, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Ki Health PARTNERS LLC DBA NEW ENGLAND INSTITUTE FOR CLINICAL RESEARCH, Stamford, Connecticut
  - Brain Matters Research, Delray Beach, Florida
  - University of Miami, Miami, Florida
  - USF Health Byrd Alzheimer's Institute, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Northern Light Acadia Hospital, Bangor, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Galen Research, Chesterfield, Missouri
  - Cleveland Clinic Lou Ruvo Center, Las Vegas, Nevada
  - Princeton Medical Institute, Princeton, New Jersey
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Department of Geriatrics, Syracuse, New York
  - James J. Peters VAMC, The Bronx, New York
  - Case Western Reserve University, Beachwood, Ohio
  - Ohio State University, Columbus, Ohio
  - Tulsa Clinical Research, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Keystone Clinical Studies, LLC, Norristown, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Geisinger Medical Clinic, Wilkes-Barre, Pennsylvania
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - CBRI, Roper Hospital, Charleston, South Carolina
  - Vanderbilt Memory & Alzheimer's Center, Nashville, Tennessee
  - The Glenn Biggs Institute for Alzheimer's and Neurodegenerative Diseases,University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Qiu Y, Jacobs DM, Messer K, Salmon DP, Wellington CL, Stukas S, Revta C, Brewer JB, Leger GC, Askew B, Donahue L, Kaplita S, Coric V, Qureshi IA, Feldman HH; Alzheimer's Disease Cooperative Study T2 Protect AD Study Group. Prognostic value of plasma biomarkers for informing clinical trial design in mild-to-moderate Alzheimer's disease. Alzheimers Res Ther. 2025 May 2;17(1):97. doi: 10.1186/s13195-025-01745-3. PMID 40317057

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 2, randomized, double-blind, placebo-controlled study was conducted in participants with mild to moderate alzheimer's disease (AD) at 44 centers in the US between 31-Jul-2018 and 23-Dec-2021.
Pre-assignment Details: A total of 687 participants were screened, of which 350 participants were randomized in a 1:1 ratio to receive troriluzole or placebo. 337 participants were not randomized due to screen failure, adverse events, lost to follow-up, withdrawal of consent, or unspecified reasons.
Groups:
- Troriluzole: Randomization phase (Randomization through Week 48): Participants received starting dose of troriluzole 140 milligrams (mg) capsules orally once daily for 2 weeks, followed by 280 mg once daily for the remaining 46 weeks of the double-blind phase.
  Open-label extension (OLE) phase (48 weeks): Participants who completed the double-blind treatment phase were offered the opportunity to enroll in an OLE phase to receive starting dose of troriluzole 140 mg capsules orally once daily for 2 weeks, followed by 280 mg orally once daily for the remaining 46 weeks.
- Placebo: Randomization phase (Randomization through Week 48): Participants received placebo matching with troriluzole for 48 weeks.
  OLE phase (48 weeks): Participants who completed the double-blind treatment phase were offered the opportunity to enroll in an OLE phase to receive starting dose of troriluzole 140 mg capsules orally once daily for 2 weeks, followed by 280 mg orally once daily for the remaining 46 weeks.
Period: Randomization Phase (Weeks 1 Through 48)
Arm/Group | Troriluzole | Placebo
Started | 178 | 172
Completed | 130 | 133
Not Completed | 48 | 39
Not completed — Withdrawal by Subject | 18 | 19
Not completed — Adverse Event | 14 | 3
Not completed — Other | 1 | 4
Not completed — Progressive disease | 3 | 2
Not completed — Lack of Efficacy | 2 | 2
Not completed — Physician Decision | 2 | 3
Not completed — Non-compliance with study drug | 4 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 2 | 3
Not completed — Death | 1 | 2
Period: OLE Phase (48 Weeks)
Arm/Group | Troriluzole | Placebo
Started | 90 (Troriluzole - Randomization Phase/ Troriluzole - OLE Phase: Participants who continued into the extension phase.) | 104 (Placebo - Randomization Phase/ Troriluzole - OLE Phase: Participants who continued into the extension phase.)
Completed | 35 | 24
Not Completed | 55 | 80
Not completed — Withdrawal by Subject | 30 | 51
Not completed — Other | 6 | 8
Not completed — Lack of Efficacy | 6 | 5
Not completed — Adverse Event | 5 | 5
Not completed — Progressive Disease | 2 | 0
Not completed — Physician Decision | 5 | 7
Not completed — Protocol Violation | 0 | 1
Not completed — Study Terminated By Sponsor | 0 | 1
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated population included enrolled and randomized participants who received at least 1 dose of blinded study therapy (troriluzole or placebo).
Groups:
- Troriluzole: Randomization phase (Randomization through Week 48): Participants received starting dose of troriluzole 140 mg capsules orally once daily for 2 weeks, followed by 280 mg once daily for the remaining 46 weeks of the double-blind phase.
  OLE phase (48 weeks): Participants who completed the double-blind treatment phase were offered the opportunity to enroll in an OLE phase to receive starting dose of troriluzole 140 mg capsules orally once daily for 2 weeks, followed by 280 mg orally once daily for the remaining 46 weeks.
- Total: Total of all reporting groups
Arm/Group | Troriluzole | Placebo | Total
Number analyzed (Participants) | 178 | 171 | 349
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (7.93) | 71.6 (7.91) | 71.7 (7.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 92 | 202
  Male | 68 | 79 | 147
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 172 | 165 | 337
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 4 | 9
  White | 170 | 163 | 333
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) Total Score at Week 48
Description: The ADAS-Cog is a structured scale that evaluates memory (word recall, word recognition), reasoning (following commands), language (naming, comprehension), orientation, ideational praxis (placing a letter in an envelope) and constructional praxis (copying geometric designs). Ratings of spoken language, language comprehension, word finding difficulty, and ability to remember test instructions were also obtained. The test was scored in terms of errors on a scale ranging from 0 (best) to 70 (worse), with higher scores indicate poorer performance and greater impairment.
Time Frame: Baseline (Day 1) and Week 48
Population: Modified Intent to Treat (mITT) population included randomized participants who received at least 1 dose of blinded study therapy (troriluzole or placebo) and who also had a baseline assessment and who have at least 1 efficacy evaluation following baseline. Participants results at Week 48 are reported.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Troriluzole: Randomization phase (Randomization through Week 48): Participants received starting dose of troriluzole 140 mg capsules orally once daily for 2 weeks, followed by 280 mg once daily for the remaining 46 weeks of the double-blind phase.
- Placebo: Randomization phase (Randomization through Week 48): Participants received placebo matching with troriluzole for 48 weeks.
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 119 | 127
units on a scale | 6.7 [5.3 to 8.1] | 6.7 [5.4 to 8.1]
Statistical Analysis 1: Comparison: Troriluzole vs Placebo; Model based summary statistics are from a mixed model with repeated measures, including fixed effects for pooled site ID, treatment, visit, treatment-by-visit interaction, baseline, baseline-by-visit interaction, mini-mental state examination (MMSE) randomization stratification, apolipoprotein E (APoE) status (carrier/non carrier), as covariates, and repeated measures for visit within participant; Test type: Superiority — Unstructure covariance structure; p = 0.9809, Mixed model with repeated measures; Least square mean difference = 0.0, 95% CI 2-sided [-1.8 to 1.8], Standard Error of Mean 0.93

2. Primary Outcome: Change From Baseline in Clinical Dementia Rating-Sum of Boxes (CDR-Sum of Boxes) Total Score at Week 48
Description: The CDR-sum of boxes is a validated composite rating of cognition and everyday functioning used in longitudinal AD research which incorporates both informant input and direct assessment of performance. It assesses through semi-structured interview 3 cognitive domains including memory, orientation, and judgement/problem solving and 3 everyday functional domains including community affairs, home and hobbies and personal care. The individual domain score ranging from 0 (none) to 3 (severe) but the scores in each of these were combined to obtain a composite score (sum of boxes) ranging from 0 (best) to 18 (worst), with higher scores indicate poorer performance and greater impairment. The individual domain scores are added to create a sum of the box scores.
Time Frame: Baseline (Day 1) and Week 48
Population: The mITT population included randomized participants who received at least 1 dose of blinded study therapy (troriluzole or placebo) and who also had a baseline assessment and who have at least 1 efficacy evaluation following baseline. Participants results at Week 48 are reported.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 118 | 127
units on a scale | 2.1 [1.7 to 2.5] | 1.9 [1.5 to 2.3]
Statistical Analysis 1: Comparison: Troriluzole vs Placebo; Model based summary statistics are from a mixed model with repeated measures, including fixed effects for pooled site ID, treatment, visit, treatment-by-visit interaction, baseline, baseline-by-visit interaction, MMSE randomization stratification, APoE status (carrier/non carrier), as covariates, and repeated measures for visit within participant; Test type: Superiority — Unstructure covariance structure; p = 0.4474, Mixed model with repeated measures; Least square mean difference = -0.2, 95% CI 2-sided [-0.8 to 0.3], Standard Error of Mean 0.28

3. Secondary Outcome: Change From Baseline in Magnetic Resonance Imaging (MRI) Hippocampal Volume at Week 48
Description: Volumetric MRI allows the in vivo assessment of brain structure volume and provides a measure of atrophy rate. Results from MRI studies suggest that the patterns of atrophy in AD, which mirror the pathological progression of the disease, can reliably be detected and tracked across time. Hippocampal volume derived from MRI correlates with histological hippocampal volume and degree of neuronal loss and AD pathology, and entorhinal cortical thickness change appears to be an early and sensitive indicator of neurodegeneration associated with AD.
Time Frame: Baseline (Day 1) and Week 48
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent deformation
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 87 | 90
percent deformation | -1.1 [-1.4 to -0.7] | -1.1 [-1.5 to -0.8]
Statistical Analysis 1: Comparison: Troriluzole vs Placebo; Model based summary statistics were from an analysis of covariance (ANCOVA) with baseline MMSE total score as covariate; Test type: Superiority — Unstructure covariance structure; p = 0.8670, ANCOVA; Least square mean difference = 0.0, 95% CI 2-sided [-0.6 to 0.5], Standard Error of Mean 0.26

4. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) Total Score at Week 48
Description: The ADCS-ADL inventory scale is validated questionnaire developed by the ADCS to assess instrumental and basic activities of daily living based on a 23-item structured interview of the AD study participant's partner. The scale ranging from 0 (none) to 78 (severe), with lower scores indicate greater impairment.
Time Frame: Baseline (Day 1) and Week 48
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 119 | 125
units on a scale | -8.9 [-10.8 to -7.1] | -7.4 [-9.2 to -5.6]
Statistical Analysis 1: Comparison: Troriluzole vs Placebo; Model based summary statistics are from a mixed model with repeated measures, including fixed effects for pooled site ID, treatment, visit, treatment-by-visit interaction, baseline, baseline-by-visit interaction, MMSE randomization stratification, APOE status (carrier/non-carrier), as covariates, and repeated measures for visit within participant; Test type: Superiority — Unstructure covariance structure; p = 0.1950, Mixed model with repeated measures; Least square mean difference = 1.6, 95% CI 2-sided [-0.8 to 3.9], Standard Error of Mean 1.21

5. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Total Score at Week 48
Description: The NPI is a well-validated, reliable, multi-item instrument to assess psychopathology in AD dementia based on the results of an interview with the study partner. The NPI evaluates both the frequency and severity of 10 neuropsychiatric features, including delusions, hallucinations, agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, irritability and lability, and aberrant motor behavior, as well as evaluates sleep and appetite/eating disorders. Frequency assessments range from 1 (occasionally, less than once per week) to 4 (very frequently, once or more per day or continuously). Severity assessments range from 1 (mild) to 3 (severe). The total score is the sum of all subscales ranging from 1 (mild) to 7 (severe), with higher scores indicate greater impairment.
Time Frame: Baseline (Day 1) and Week 48
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 120 | 125
units on a scale | 2.3 [0.2 to 4.4] | 3.8 [1.8 to 5.8]
Statistical Analysis 1: Comparison: Troriluzole vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — Unstructure covariance structure; p = 0.2583, Mixed model with repeated measures; Least square mean difference = 1.5, 95% CI 2-sided [-1.1 to 4.1], Standard Error of Mean 1.31

6. Secondary Outcome: Change From Baseline in Mini-Mental Status Examination (MMSE) Total Score at Week 48
Description: The MMSE is a frequently used screening instrument for AD drug studies. It evaluates orientation, memory, attention, concentration, naming, repetition, comprehension, and ability to create a sentence and to copy 2 intersecting pentagons. The MMSE scale ranging from 0 (worse) to 30 (best), with a lower score indicate more cognitive impairment.
Time Frame: Baseline (Day 1) and Week 48
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 121 | 128
units on a scale | -3.6 [-4.4 to -2.9] | -3.2 [-4.0 to -2.5]
Statistical Analysis 1: Comparison: Troriluzole vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — Unstructure covariance structure; p = 0.4191, Mixed model with repeated measures; Least square mean difference = 0.4, 95% CI 2-sided [-0.6 to 1.3], Standard Error of Mean 0.48

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in participants or clinical investigation participants administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. A serious AE (SAE) is defined as any event that met any of the following criteria at any dose: death; life-threatening; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect in the offspring of a participant who received study drug; other important medical events that may have jeopardized the participant and may have required medical or surgical intervention to prevent one of the other serious outcomes. An AE is considered "Related" for causality designations of possible, probable and definite.
Time Frame: TEAEs were reported from first dose of study drug up to end of study treatment, maximum of 96 weeks.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Troriluzole - Randomization Phase: Participants received starting dose of troriluzole 140 mg capsules orally once daily for 2 weeks, followed by 280 mg once daily for the remaining 46 weeks of the double-blind phase.
- Placebo - Randomization Phase: Participants received placebo matching with troriluzole for 48 weeks.
- Troriluzole - Randomization Phase/ Troriluzole - OLE Phase; Placebo - Randomization Phase/ Troriluzole - OLE Phase: Participants who completed the double-blind treatment phase were offered the opportunity to enroll in an OLE phase to receive starting dose of troriluzole 140 mg capsules orally once daily for 2 weeks, followed by 280 mg orally once daily for the remaining 46 weeks.
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase | Troriluzole - Randomization Phase/ Troriluzole - OLE Phase | Placebo - Randomization Phase/ Troriluzole - OLE Phase
Number analyzed (Participants) | 178 | 171 | 90 | 103
Participants
  Any TEAEs | 146 | 116 | 57 | 66
  Any serious TEAEs | 24 | 14 | 9 | 16
  Any fatal AE | 2 | 2 | 0 | 2
  Any serious TEAEs considered related | 3 | 1 | 0 | 3
  Drug withdrawn due to an TEAE | 16 | 3 | 5 | 12

8. Other Pre Specified Outcome: Change From Baseline in Magnetic Resonance Imaging (MRI) Hippocampal Volume at Week 48 in Mild Subgroup
Description: Subgroup of participants MMSE Category = Mild. The MMSE scale ranging from 0 (worse) to 30 (best), with a lower score indicating more cognitive impairment. Mild are participants with a baseline MMSE score greater than or equal to 20.
Time Frame: Baseline (Day 1) and Week 48
Measure: Least Squares Mean (95% Confidence Interval); unit: percent deformation
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 48 | 49
percent deformation | -1.1 [-1.6 to -0.6] | -1.6 [-2.1 to -1.0]
Statistical Analysis 1: Comparison: Troriluzole vs Placebo; Model based summary statistics are from an ANCOVA with baseline MMSE total score as covariate; Test type: Superiority; p = 0.2240, ANCOVA; Least square mean difference = -0.5, 95% CI 2-sided [-1.2 to 0.3], Standard Error of Mean 0.38

9. Post Hoc Outcome: Number of Responders in Participants With ADAS-cog Total Change and MRI Hippocampal Volume Change at Week 48 in Mild APOE e4 Carrier Subgroup
Description: Mild APOE e4 carrier subgroup are participants with a baseline MMSE score greater than or equal to 20 with APOE e4 genotype. Responder based on ADAS-cog Total Change less than or equal to 1 and MRI Hippocampal Volume Change greater than or equal to -2.09. ADAS-cog change and MRI Hippcampal volume change criteria based on 25th percentile.
Time Frame: Baseline (Day 1) and Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Troriluzole | Placebo
Number analyzed (Participants) | 45 | 44
Participants | 14 | 4
Statistical Analysis 1: Comparison: Troriluzole vs Placebo; Test type: Superiority; p = 0.0161, Fisher Exact

ADVERSE EVENTS:
Time Frame: TEAEs were reported from first dose of study drug up to end of study treatment, maximum of 96 weeks.
Description: Treated population included enrolled and randomized participants who received at least 1 dose of blinded study therapy (troriluzole or placebo).
Arm/Group | Troriluzole - Randomization Phase | Placebo - Randomization Phase | Troriluzole - Randomization Phase/ Troriluzole - OLE Phase | Placebo - Randomization Phase/ Troriluzole - OLE Phase
All-Cause Mortality (participants affected / at risk) | 2/178 | 2/171 | 0/90 | 2/103
Serious Adverse Events (participants affected / at risk) | 24/178 | 14/171 | 9/90 | 16/103
Other Adverse Events (participants affected / at risk) | 81/178 | 53/171 | 29/90 | 31/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Troriluzole - Randomization Phase (N=178) | Placebo - Randomization Phase (N=171) | Troriluzole - Randomization Phase/ Troriluzole - OLE Phase (N=90) | Placebo - Randomization Phase/ Troriluzole - OLE Phase (N=103)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0
Hypothermia (General disorders) | 1 | 0 | 0 | 0
Pelvic mass (General disorders) | 1 | 0 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 1 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Colonic abscess (Infections and infestations) | 1 | 0 | 1 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 1 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0
Frostbite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Embolic cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropsychiatric symptoms (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Paranoia (Psychiatric disorders) | 1 | 0 | 0 | 0
Somnambulism (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Troriluzole - Randomization Phase (N=178) | Placebo - Randomization Phase (N=171) | Troriluzole - Randomization Phase/ Troriluzole - OLE Phase (N=90) | Placebo - Randomization Phase/ Troriluzole - OLE Phase (N=103)
Diarrhoea (Gastrointestinal disorders) | 15 | 6 | 1 | 3
Oedema peripheral (General disorders) | 9 | 2 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 5 | 1
Urinary tract infection (Infections and infestations) | 15 | 12 | 5 | 5
Fall (Injury, poisoning and procedural complications) | 19 | 11 | 10 | 7
Liver function test increased (Investigations) | 5 | 0 | 2 | 6
Weight decreased (Investigations) | 16 | 4 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 16 | 2 | 1 | 1
Dizziness (Nervous system disorders) | 10 | 13 | 3 | 2
Headache (Nervous system disorders) | 6 | 14 | 3 | 3
Anxiety (Psychiatric disorders) | 9 | 7 | 3 | 3

LIMITATIONS AND CAVEATS:
All participants in the OLE phase underwent a termination visit 2 weeks after the last dose of troriluzole.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-09-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT03605667/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT03605667/SAP_001.pdf